CLINICAL TRIAL: NCT03980171
Title: A Multicenter, Open Label, Phase Ib/II Study of Lenalidomide, Venetoclax and Obinutuzumab in Patients With Treatment-Naïve Follicular Lymphoma
Brief Title: Study of Lenalidomide, Venetoclax and Obinutuzumab in Patients With Treatment-Naïve Follicular Lymphoma
Acronym: LEVERAGE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/45
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab; venetoclax; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obinutuzumab+venetoclax+lenalidomide (Experimental): Patients in both dose escalation and dose expansion will receive 6 cycles of induction treatment consisting of obinutuzumab (flat dose of 1000mg) and protocol defined dose levels of venetoclax and lenalidomide.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Lenalidomide

INTERVENTIONS:
Drug: Obinutuzumab — A flat dose of 1000mg IV will be given every cycle during induction. a cycle is 28 days.During maintenance 1000mg IV will be given every second cycle for upto 2 years.
  Other Names: GAZYVA; GAZYVARO
Drug: Venetoclax — During dose escalation, the doses for venetoclax can be 400mg daily days 1-10, 800mg daily days 1-10, 400mg daily continuous or 800mg daily continuous. 6 cycles of treatment will be given during induction. Once the recommended phase 2 dose (RP2D) is established that dose will be used in dose expansion. A further 6 cycles of venetoclax will be given during maintenance if required based on response at the end of induction.
  Other Names: ABT-199 (A-1195425.0); Venclexta; Venclyxto
Drug: Lenalidomide — During dose escalation, the doses of lenalidomide can be 15mg for days 1-21 or 20mg for days 1-21. 6 cycles of treatment will be given during induction. During maintenance the dose of lenalidomide will be 10mg continuous for a further 6 cycles if required based on response at the end of induction.
  Other Names: Revlimid

SUMMARY:
The trial will investigate the combination of venetoclax, obinutuzumab and lenalidomide in patients with treatment-naïve follicular lymphoma. Patients will receive induction treatment for 0.5 years with venetoclax, obinutuzumab and lenalidomide followed by maintenance treatment for upto 2 years. Maintenance treatment will be determined by the response at the end of induction. Following completion of treatment patients will be followed up for 3 years after the last patient completes induction treatment.

DETAILED DESCRIPTION:
This is a phase Ib/II (dose escalation/dose expansion), single-arm multi-centre clinical trial of venetoclax plus obinutuzumab and lenalinomide in patients with treatment-naïve follicular lymphoma. The trial involves an initial dose escalation phase followed by an expansion phase. Patients in both the dose escalation and expansion phases will receive 6 cycles of induction treatment. After patients finish induction treatment, they will undergo PET-CT scan, the results of which will determine further therapy. Patients in CR or SD/PR from the PET-CT scan result will receive up to 2 years of maintenance therapy. Patients in PD from the PET-CT result will not receive any further study treatment. All patients will be followed up for 3 years after the last patient has completed induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent.
2. Patient has histologically confirmed follicular lymphoma WHO grade 1-3A and non-contiguous or bulky (>7cm) stage II and stage III or IV according to Lugano criteria 2014, irrespective of FLIPI score
3. Patient meets ≥1 Groupe d'Etude des Lymphomes Folliculaires (GELF) criterion for treatment.
4. Bi-dimensionally measurable disease, with at least one mass lesion ≥ 2 cm in longest diameter.
5. Male or female age ≥ 18 years at signing consent
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Adequate organ and haematologic function within 10 days prior to registration, defined by:

   * Haemoglobin ≥80g/L
   * ANC ≥1 x 109/L and platelet count ≥75 x 109/L; unless due to marrow infiltration or hypersplenism (in which case ANC ≥ 0.5 x 109/L and platelets ≥ 50 x 109/L)
   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) <2.5 x upper limit of normal (ULN)
   * International normalized ratio >1.5 x ULN for patients not receiving therapeutic anticoagulation
   * Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤1.5 x ULN unless due to the presence of an inhibitor (e.g. lupus anticoagulant)
   * Bilirubin <2.0 x ULN unless due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin
   * Creatinine clearance ≥50ml/min(Cockcroft-Gault)
8. Able to comply with protocol requirements and follow-up procedures.
9. Female patients of childbearing potential (FCBP) must be willing to use two methods of birth control simultaneously or be surgically sterile, or abstain from heterosexual activity for at least 28 days before starting lenalidomide and for the course of the study through to 18 months after the last dose of obinutuzumab, 28 days after the last dose of lenalidomide and 30 days after the last dose of venetoclax, whichever is longer. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 24 consecutive months (Refer to Appendix 4).
10. Sexually active males must agree to use a condom during sexual contact with a pregnant female or a female of child-bearing potential (FCBP) for the course of the study through to 18 months after the last dose of obinutuzumab, 28 days after the last dose of lenalidomide and 30 days after the last dose of venetoclax, whichever is longer, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. WHO grade 3B follicular lymphoma, biopsy proven or clinically suspected histologic transformation to diffuse large B-cell lymphoma
2. Known central nervous system lymphoma or leptomeningeal disease.
3. History of other malignancy that could affect compliance with the protocol or interpretation of results Patients with a history of curatively treated basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible.

   Patients with a malignancy that has been treated with curative intent may be included provided they remain in remission without treatment for ≥ 2 years prior to enrollment
4. Has had prior systemic therapy for follicular lymphoma (with the exception of corticosteroid monotherapy to control disease related symptoms).
5. Major surgery or a wound that has not fully healed within 4 weeks prior to registration.
6. Patient is unable to swallow tablets.
7. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of venetoclax or lenalidomide capsules, or put the study outcomes at undue risk.
8. Known hypersensitivity to any of the study drugs or their components (obinutuzumab, L-histidine, L-histidine hydrochloride monohydrate, Trehalose dehydrate, Poloxamer 188), humanized or murine monoclonal antibodies, xanthine oxidase inhibitors or rasburicase.
9. Has received the following agents within 7 days prior to registration:

   * Steroid therapy with anti-neoplastic intent (with the exception of ≤7 days of prednisolone or equivalent at doses of ≤100mg daily to control lymphoma symptoms prior to cycle 1 day 1)
   * Strong CYP3A inhibitors (See section 7.10.3)
   * Strong CYP3A inducers (See section 7.10.3)
   * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days of registration
10. Has a history of stroke or intracranial hemorrhage within 6 months prior to registration.
11. Has a known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment.
12. Requires the use of vitamin K antagonists (because of potential drug-drug interactions that may potentially increase the exposure of warfarin).
13. Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody.

    Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to receive prophylactic lamivudine or entecavir and undergo monthly DNA testing during (and for 6 months following completion of) treatment.
14. Receipt of live-virus vaccines within 28 days prior to registration or need for live-virus vaccines at any time during study treatment.
15. Pregnant or lactating, or intending to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | During the first 2 cycles of induction during dose escalation which is expected to be completed in 1.5 years.
  A toxicity that prevents further administration of the trial treatment at that dose level.
Recommended phase II dose (RP2D) of venetoclax in combination with lenalidomide and obinutuzumab | During dose escalation (1.5 years)
  The highest dose level at which the incidence of DLT was less than 2/6
Complete response (CR) at the end of induction | 3.5 years from first patient commencing treatment
  Investigator assessed CR rate by PET-CT after induction (end of cycle 6) by 2014 Lugano criteria
Adverse events (AEs) of venetoclax, lenalidomide and obinutuzumab | From signing consent until after completion of study treatment (6.75 years)
  Type, grade and relationship to treatment of AEs, assessed according to Common Terminology of Coding of Adverse Events (CTCAE) v5.0.
Rate of treatment-emergent AEs that require discontinuation or dose modification of study drug | From signing consent until after completion of study treatment (6.75 years)
  Type and grade of treatment-emergent AEs, assessed according to CTCAE v5.0, requiring discontinuation of study drug or dose reductions or interruptions
Overall response rate (ORR) | 3.5 years from first patient commencing treatment
  Investigator assessed ORR (complete response (CR) or partial response (PR)) by PET-CT assessed by 2014 Lugano criteria after 6 cycles of induction treatment (0.5 years)
CR at 2.5 years from commencement of induction treatment | 5.5 years from first patient commencing treatment
  CR based on 2014 Lugano criteria
Progression free survival (PFS) | From commencement of treatment to end of study (6.75 years)
  PFS will be defined as the time from enrolment date to the first date of objectively documented progressive disease (PD) or date of death from any cause. Patients without documented progressive disease and who have not died by the end of the study will be censored at the date of last disease assessment.
Duration of response (DOR) | From commencement of treatment to end of study (6.75 years)
  DOR will be measured in the subset of patients who achieved CR or PR and it is defined as the time from the first documented disease response to the earliest recurrence or progressive disease. Deceased patients without recurrence or progressive disease will be censored at the date of death.
Time to next anti-lymphoma treatment (TTNT) | From commencement of treatment to end of study (6.75 years)
  TTNT will be measured from enrolment date to date of initiation of next anti-cancer therapy (for follicular lymphoma) or date of death from any cause. Patients who do not start next anti-cancer therapy by the end of the study will be censored at the date of last contact.
Overall survival (OS) | From commencement of treatment to end of study (6.75 years)
  OS will be measured from enrolment date to the date of death from any cause. Patients who have not died by the study close-out date will be censored at their last visit date. Patients who are lost to follow-up before the close-out date and who are not known to have died will be censored at the date they were last known to be alive.
Quality of life (QoL) | From commencement of treatment to end of treatment (5.5 years)
  QoL will be measured using Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym).
  The FACT-Lym is a disease-specific 42-item questionnaire that has been validated for the purpose of assessing health-related quality of life (HRQoL) in patients with various forms of lymphoma.The FACT-Lym consists of FACT-G subscales: Physical Well-Being (7 items), Social/Family Well-Being (7 items), Emotional Well-Being (6 items), Functional Well-Being (7 items), and the Lymphoma subscale: Additional Concerns (15 items). FACT-Lym questions are scored on a 5-point Likert scale from 0 to 4 (0 being not at all and 4 being very much).

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Townsville Hospital and Health Services, Townsville, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No